CLINICAL TRIAL: NCT03826056
Title: Neurology Inpatient Clinical Education Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Vijay Renga, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: D19046
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-01

CONDITIONS: Myasthenia Gravis; Guillain-Barre Syndrome; Multiple Sclerosis; Seizures; Parkinsonism; Meningitis; Encephalitis; Headache; Vestibular Disorder; Spondylosis; Normal Pressure Hydrocephalus
Keywords: clinical education
MeSH Terms: conditions — Myasthenia Gravis; Guillain-Barre Syndrome; Multiple Sclerosis; Seizures; Parkinsonian Disorders; Meningitis; Encephalitis; Headache; Vestibular Diseases; Spondylosis; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Intervention Model Description: Study team members will randomize patients to receive either the current standard hospital education material or the new personalized education material. Investigators will use a stratified randomization process to allocate the patients from different categories including age range, gender, and discharge diagnosis into each group. Thereby the investigators will achieve equal distribution of diagnoses and other demographics among groups in real time. They will review the two groups when performing statistical analysis near the end of the study to ensure heterogeneity of distribution.
  A study team member who has also been a member of the care team will use the either the current hospital standard or the new personalized education materials to explain the discharge diagnosis to the patient, the treatment, and the follow up needed. The study team member will also give a survey with a preaddressed envelope to each participant to complete at his or her convenience.
Who Masked: Participant
Masking Description: The patient will not be informed of whether he or she is receiving the current hospital standard or the new personalized patient education intervention. The study team member will known which intervention is being used for patient education. The intervention arm will not be blinded in the data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current standard education group (Active Comparator): A study team member will use the current hospital standard educational material to explain the discharge diagnosis to the patient, the treatment, and the follow up needed. The study team member will also give a survey with a preaddressed envelope to each participant to complete at his or her convenience.
  Interventions: Behavioral: Current standard discharge educational intervention
- New personalized education group (Experimental): A study team member will use the new personalized educational materials to explain the discharge diagnosis to the patient, the treatment, and the follow up needed. The study team member will also give a survey with a preaddressed envelope to each participant to complete at his or her convenience.
  Interventions: Behavioral: Personalized discharge educational intervention

INTERVENTIONS:
Behavioral: Current standard discharge educational intervention — The patients will receive the current hospital standard discharge educational material which explains the diagnosis, new medications, follow up and any activity/diet restrictions. A member of the study team will explain this material to the patient and answer any questions.
  Arms: Current standard education group
Behavioral: Personalized discharge educational intervention — The patients will receive a new personalized discharge educational material which will explain the specifics of their disorder, the treatment, and prognosis. The materials will contain simple, organized explanations and graphics. A member of the study team will explain this material to the patient and answer any questions.
  Arms: New personalized education group

SUMMARY:
The objective of this study is to compare the effectiveness of a personalized patient education program to the current hospital education and evaluate its impact using patient satisfaction scores.

The investigators hypothesize that a personalized patient education intervention will increase patient's understanding of their diagnosis and satisfaction with the care as reflected in the survey results.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Must have the capacity to consent and understand the study related activities and education materials.

Exclusion Criteria:

* Under the age of 18
* Have a condition that impairs the ability to understand the study, its risks, and appropriately consent for the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction scores | Subjects will be expected to mail the feedback forms within 2 weeks of discharge. Investigators will mail a single reminder prepaid return mail with a copy of the questionnaire to patients who do not respond within this time allowing 1 month total time.
  The patients will answer a survey consisting of seven multiple-choice questions regarding their perception of the education intervention. Each questions will be scored on a scale of one to four for a total possible score of 28 for all 7 questions. A score of 1 indicates a negative perception of the education whereas 4 indicates the most positive impression. Therefore the lowest possible score is 7 for a severely negative perception of the education and the highest score is 28 for a very positive impression of the education program. Only the total scores will be compared for statistical analysis. Scores from patients in the current standard and new personalized education intervention groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Renga, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth- Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Investigators will protect patients' identity by using identification numbers that do not correspond to any personal identification information. They will enter the survey results to the institution's safely encrypted database.